CLINICAL TRIAL: NCT02036879
Title: Gender Disparity and Hormones in Cystic Fibrosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Raksha Jain, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU 072013-079
Record Dates: First submitted 2013-12-26; First posted 2014-01-15 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Cystic Fibrosis (CF)
Keywords: Cystic Fibrosis; Loestrin; Hormone
MeSH Terms: conditions — Cystic Fibrosis | interventions — norethindrone acetate, ethinyl estradiol, ferrous fumarate drug combination; Norethindrone Acetate; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Main study (No Intervention): The main study is an observational study.
  All women will be followed for one menstrual cycle (or approximately one month) observationally off of any hormone supplementation. They will have 3 study visits corresponding to their menstrual cycle phases (menses, ovulation, and luteal).
  Women participating in the main study may participate in the optional interventional sub-study.
  Men participating in this study will be followed for 1 month observationally. They will have 3 study visits that correlate with the female arm of this study.
- Loestrin Optional Substudy (Experimental): Women participating in the main study may participate in the optional sub-study. Following a negative urine pregnancy test, women will be started on once daily oral Loestrin (1.5 mg norethindrone + 0.03 mg ethyl estradiol). They will be followed for two months on this agent and have 2 additional study visits.
  Interventions: Drug: Loestrin (norethindrone acetate and ethinyl estradiol)

INTERVENTIONS:
Drug: Loestrin (norethindrone acetate and ethinyl estradiol) — This is an optional substudy that females participating in the main study can choose to participate in. Loestrin, an oral contraceptive or birth control pill, will be prescribed and taken daily for approximately 2 months.
  Arms: Loestrin Optional Substudy

SUMMARY:
The objective of this study is to investigate the impact of hormones on lung disease in Cystic Fibrosis (CF) patients. Due to improved therapies, CF patients are living longer and healthier lives than they did 20 years ago. However, females have been shown to have a survival disadvantage. The median life expectancy is 33 in women and 37 in men with CF. The hypothesis is that estrogen and/or progesterone negatively impact lung health in CF. Therefore, understanding the impact of sex hormones (including the use of birth control pills) on the disease process is increasingly important. The purpose of this study is to determine if lung function, respiratory symptoms, or various markers of lung health change during different phases of the natural ovulatory cycle in order to understand if estrogen or progesterone hormones are impacting the disease relative to fluctuations in men with stable testosterone levels. The research objectives of this project are to:

* Determine if lung function, respiratory symptoms, or various markers of lung health change during different hormonal phases of the ovulatory cycle in women.
* Determine if men change lung function, respiratory symptoms, or various markers of lung health over time.
* Determine if oral contraceptive pills in women stabilize fluctuations in symptoms and improve lung health.

ELIGIBILITY:
Inclusion Criteria:

* Male and female cystic fibrosis patients
* Must be greater than or equal to 18 years of age.
* All subjects must understand and sign the informed consent.
* Subjects must have the ability to read and write in English.
* Female subjects starting this study must be willing to use a double barrier method of birth control (such as condom or diaphragm) used with a spermicide (a substance that kills sperm), while participating in the study.

Exclusion Criteria for Main Study:

* Women who are pregnant, breast feeding, or who have had an oophorectomy.
* Women who have received a hormone contraceptive injection (such as Depo Provera) within the last 3 months.

Exclusion Criteria for Substudy:

* Men
* Women who have a history of breast cancer, abnormal vaginal bleeding, liver disease, coronary artery disease, cerebrovascular disease, uncontrolled hypertension, diabetes mellitus with vascular disease, or have had a stroke, heart attack, or blood clot within the past year, due to a possible reaction to Loestrin.
* Women who currently smoke cigarettes, due to the increased risk of serious cardiovascular events with Loestrin use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in percent predicted forced expiratory volume in 1 second (FEV1) | Through Visit 5, if applicable (or approximately 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Raksha Jain, MD, MSCI, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Children's Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas